CLINICAL TRIAL: NCT02083354
Title: An Open-Label, Multi-Center Study to Investigate the Objective Response Rate of Dabrafenib in Combination With Trametinib in Subjects With BRAF V600 Mutation-Positive Melanoma
Brief Title: Study to Investigate the Objective Response Rate of Dabrafenib in Combination With Trametinib in Subjects With BRAF V600 Mutation-Positive Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200104; CDRB436B2205 (Other: Novartis)
Record Dates: First submitted 2014-02-13; First posted 2014-03-11 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cancer; Melanoma
Keywords: melanoma; dabrafenib; trametinib; malignant skin cancer; skin cancer; BRAF V600 Mutation-Positive Melanoma
MeSH Terms: conditions — Neoplasms; Melanoma; Skin Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): All subjects will receive the combination of dabrafenib (150 mg) and trametinib (2 mg) in the morning at approximately the same time every day. The second dose of dabrafenib (150 mg) alone will be administered approximately 12 hours after the morning dose. Subjects will continue study treatment until disease progression, death, unacceptable toxicity, withdrawal of consent, or study closure
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib will be provided as 50 mg and 75 mg capsules. Each capsule will contain 50 mg or 75 mg of free base (present as the mesylate salt)
Drug: Trametinib — Trametinib study medication will be provided as 0.5 mg and 2.0 mg tablets. Each tablet will contain 0.5 mg or 2.0 mg of trametinib parent (present as the DMSO solvate)

SUMMARY:
This was a single-arm, open-label, multi-center, Phase II study to evaluate dabrafenib and trametinib combination therapy in subjects with BRAF V600 mutation-positive, unresectable or metastatic Acral lentiginous or cutaneous melanoma. This study evaluated the objective response rate (ORR), progression free survival (PFS), duration of response, overall survival (OS), safety and efficacy, to assess steady state (all subjects) exposure to dabrafenib, dabrafenib metabolites, and trametinib and characterize the population pharmacokinetics (PK) and pharmacodynamics (PD) of dabrafenib and trametinib. Enrolled subjects were administered dabrafenib 150 milligram (mg) orally twice daily and trametinib 2 mg orally once daily. Treatment continued until disease progression, death, unacceptable toxicity, or withdrawal of consent, or study closure. After treatment discontinuation, subjects were followed for survival and disease progression as applicable.

DETAILED DESCRIPTION:
This was an open-label, single arm, Phase IIA, multi-center study to evaluate the Objective response rate (ORR) of dabrafenib and trametinib combination therapy in East Asian subjects that have BRAF V600 mutationpositive Stage IIIC (unresectable) or Stage IV (metastatic) acral lentiginous melanoma (ALM) or cutaneous melanoma.

All subjects enrolled received oral dabrafenib 150 mg bid in combination with oral trametinib 2 mg once daily. A primary analysis presented the efficacy, safety and pharmacokinetics (PK) data up to the data cut-off date of 23-Feb-2018. Based on these results, dabrafenib and trametinib combination was approved in the People's Republic of China (PRC) for the treatment of BRAF-mutation positive unresectable or metastatic melanoma. Data from Mainland Chinese subjects from 01-Jul-2019 onwards are not included due to local regulations in China.

Subjects continued study treatment until disease progression, death, unacceptable toxicity, withdrawal of consent, or study completion. After treatment discontinuation, subjects went into follow-up for survival and disease progression as applicable. Subjects could continue study treatment after disease progression if they achieved clinical response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 or stable disease with tumour reduction; had no overt signs of toxicity; had Eastern Cooperative Oncology Group (ECOG) performance status of ≤1 and did not require immediate surgical or radiological intervention.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* >=18 years of age.
* Histologically confirmed acral lentiginous or cutaneous melanoma that is either Stage IIIC (unresectable) or Stage IV (metastatic), and BRAF V600 mutation-positive. The test was to have been conducted at a designated central laboratory.
* Measurable disease (i.e., present with at least one measurable lesion) by RECIST version1.1.
* Performance status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values) must be <=Grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.0) at the time of enrolment.
* Able to swallow and retain oral medication and must not have had any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Women of child-bearing potential must have had a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, from 14 days prior to enrolment, throughout the treatment period and for 4 months after the last dose of study treatment.
* Adequate baseline organ function as defined below: Absolute Neutrophil Count:>= 1.2 × 10^9/liter (L); Hemoglobin: >=9 grams (g)/deciliter (dL); Platelet count: >=100 x 10^9/L; Prothrombin Time/International Normalized Ratio (INR) (Subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to enrolment) and Partial Thromboplastin Time: <=1.5 x Upper Limit of Normal (ULN); Albumin: >=2.5 g/dL; Total bilirubin: <=1.5 x ULN; Aspartate aminotransferase and Alanine aminotransferase: <=2.5 x ULN; Calculated creatinine clearance (Calculate creatinine clearance using standard Cockcroft-Gault formula): >=50 milliliter (mL)/ minute (min); Left Ventricular Ejection Fraction (LVEF) (ECHO scans must be used throughout the study) : >= Lower limit of normal (LLN) by ECHO.
* Subjects with East Asian origin.

Exclusion Criteria:

* Primary mucosal or ocular melanoma.
* Prior treatment with a BRAF inhibitor (including but not limited to dabrafenib, vemurafenib, LGX818, and XL281/BMS-908662) or a MEK inhibitor (including but not limited to trametinib, AZD6244, and RDEA119).
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic anti-cancer therapy, or immuno anti-cancer therapy within 21 days prior to enrolment /or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrolment. (Note: Ipilimumab, pembrolizumab and nivolumab treatment must ended at least 8 weeks prior to enrollment).
* Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to enrolment. (Note: in case ipilimuamb, pembrolizmab and nivolumab are investigational drug in the regions and countries, and in case of PD-L1 antibody, these investigational treatment must have ended at least 8 weeks prior to enrollment ).
* Current use of a prohibited medication.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* A history of Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and/or HCV will be permitted).
* Leptomeningeal or brain metastases or metastases causing spinal cord compression that were: symptomatic or untreated or not stable for 3 months (must be documented by imaging) or requiring corticosteroids. Subjects that were on a stable dose of corticosteroids >1 month or on replacement dose only, or have been off of corticosteroids for at least 2 weeks can be enrolled with approval of the medical monitor. Subjects must also have been off of enzyme-inducing anticonvulsants for >4 weeks.
* History of malignancy other than disease under study within 3 years of study enrolment with exceptions of subjects with a history of completely resected non-melanoma skin cancer, or subjects with indolent second malignancies were eligible only after the approval of the sponsor's medical monitor.
* History of malignancy with confirmed activating RAS mutation at any time. Note: Prospective RAS testing was not required. However, if the results of previous RAS testing were known, they must have been used in assessing eligibility
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could have interfered with the subject's safety, obtaining informed consent, or compliance with study procedures.
* A history or evidence of cardiovascular risk including any of the following: Current LVEF < Institutional LLN; A QTc interval corrected for heart rate >=480 millisecond (msec) (using Bazett's formula); A history or evidence of current clinically significant uncontrolled arrhythmias. Clarification: Subjects with atrial fibrillation controlled for >30 days prior to dosing are eligible; A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization; A history or evidence of current >=Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines; Patients with intra-cardiac defibrillators; Treatment refractory hypertension defined as a blood pressure of systolic >140 millimeters of mercury (mmHg) and/or diastolic >90 mmHg which cannot be controlled by anti-hypertensive therapy; Known cardiac metastases; Abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not have been entered in study.
* Uncorrectable electrolyte abnormalities (e.g. hypokalaemia, hypomagnesaemia, hypocalcaemia determined by blood chemistry), long QT syndrome or taking medicinal products known to prolong the QT interval.
* A history or current evidence of retinal vein occlusion (RVO) .
* Pregnant or nursing females.
* History of or current diagnosis of interstitial lung disease or pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- China (4):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Tuenmen, Hong Kong
- Novartis Investigative Site, Seoul, South Korea
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mao L, Ding Y, Bai X, Sheng X, Dai J, Chi Z, Cui C, Kong Y, Fan Y, Xu Y, Wang X, Tang B, Lian B, Yan X, Li S, Zhou L, Wei X, Li C, Guo J, Zhang X, Si L. Overall Survival of Patients With Unresectable or Metastatic BRAF V600-Mutant Acral/Cutaneous Melanoma Administered Dabrafenib Plus Trametinib: Long-Term Follow-Up of a Multicenter, Single-Arm Phase IIa Trial. Front Oncol. 2021 Aug 24;11:720044. doi: 10.3389/fonc.2021.720044. eCollection 2021. PMID 34504796
- [Derived] Si L, Zhang X, Shin SJ, Fan Y, Lin CC, Kim TM, Dechaphunkul A, Maneechavakajorn J, Wong CS, Ilankumaran P, Lee DY, Gasal E, Li H, Guo J. Open-label, phase IIa study of dabrafenib plus trametinib in East Asian patients with advanced BRAF V600-mutant cutaneous melanoma. Eur J Cancer. 2020 Aug;135:31-38. doi: 10.1016/j.ejca.2020.04.044. Epub 2020 Jun 10. PMID 32534242

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 77 participants were enrolled in the study.
Groups:
- Arm 1: All subjects received the combination of dabrafenib (150 mg) and trametinib (2 mg) in the morning at approximately the same time every day. The second dose of dabrafenib (150 mg) alone was to be administered approximately 12 hours after the morning dose. Subjects were to continue study treatment until disease progression, death, unacceptable toxicity, withdrawal of consent, or study closure
Period: Overall Study
Arm/Group | Arm 1
Started | 77
Completed (These subjects show as ongoing in the clinical database even though no subjects are currently ongoing, as no changes to the data were permitted after 30-Jun-2019 due to local regulations in China.) | 13
Not Completed | 64
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 3
Not completed — Disease progression | 46
Not completed — Study closed/terminated | 5

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 77
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: To determine ORR of dabrafenib in combination with trametinib in subjects with BRAF V600 mutation-positive, unresectable or metastatic melanoma. ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 and as assessed by the investigator.
Time Frame: Up to 35 months
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 77
Percentage of Participants | 61 [49.2 to 72.0]

2. Secondary Outcome: Progression-free Survival (PFS) - Median
Description: PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause
Time Frame: Up to 36 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 77
months | 9.17 [7.26 to 12.88]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
  Censored, follow-up ongoing - These subjects show as ongoing in the clinical database even though no subjects are currently ongoing, as no changes to the data were permitted after 30-Jun-2019 due to local regulations in China.
Time Frame: Up to 36 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 77
Participants
  Progressive Disease (PD) (event) | 52
  Died (event) | 4
  Censored, follow-up ended | 10
  Censored, follow-up ongoing | 11

4. Secondary Outcome: Duration of Response (DOR) - Estimate for Duration of Response - Median
Description: Duration of response is defined as the time from first documented evidence of complete response (CR) or partial response (PR) until the earliest date of documented radiological progression or death due to any cause among subjects who achieved a confirmed CR or PR.
Time Frame: Up to 36 months
Population: Full analysis set, for participants who achieved CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1
Number analyzed (Participants) | 48
Months | 12.65 [5.62 to 25.23]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time from first documented evidence of complete response (CR) or partial response (PR) until the earliest date of documented radiological progression or death due to any cause among subjects who achieved a confirmed CR or PR.
  Censored, follow-up ongoing - These subjects show as ongoing in the clinical database even though no subjects are currently ongoing, as no changes to the data were permitted after 30-Jun-2019 due to local regulations in China.
Time Frame: Up to 36 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
Participants
  PFS - Disease Progression | 27
  PFS - Death | 2
  PFS - Censored, follow-up ended | 9
  PFS - Censored, follow-up ongoing | 10

6. Secondary Outcome: Overall Survival (OS) - Median
Description: OS is defined as the interval from first dose of study treatment to the date of death, irrespective of the cause of death; subjects still alive will be censored at the date of the last contact
Time Frame: Approximately 5 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1
Number analyzed (Participants) | 77
Months | 22.90 [16.62 to 27.40]

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval from first dose of study treatment to the date of death, irrespective of the cause of death; subjects still alive will be censored at the date of the last contact.
  Censored, follow-up ongoing - These subjects show as ongoing in the clinical database even though no subjects are currently ongoing, as no changes to the data were permitted after 30-Jun-2019 due to local regulations in China.
Time Frame: Approximately 5 years
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 77
Participants
  Died (Event) | 43
  Censored, follow-up ended | 13
  Censored, follow-up ongoing | 21

8. Secondary Outcome: Number of Participants With Adverse Events
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 51 months (for both dabrafenib and also Rametinib).
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 77
Participants
  Adverse events - all grades | 76
  Adverse events - Treatment-related - all grades | 69
  SAEs - all grades | 18
  SAEs - Treatment-related - all grades | 9
  Fatal SAEs - all grades | 4
  Fatal SAEs - Treatment-related - all grades | 1
  AEs leading to discontinuation - all grades | 6
  AEs leading to discontinuation - Treatment-related - all grades | 3
  AEs leading to dose adjustment/interruption - all grades | 39
  AEs leading to dose reduction - all grades | 23

9. Secondary Outcome: Population Pharmacokinetics of Dabrafenib - Cmax
Description: Cmax is the maximum peak concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 2950 (72.8)
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 2300 (70.6)

10. Secondary Outcome: Population Pharmacokinetics of Dabrafenib - Tmax
Description: Tmax is Time to Cmax (maximum peak concentration).
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Median (Full Range); unit: hr
Arm/Group | Arm 1
Number analyzed (Participants) | 20
hr
  Day 1 | 1.95 [0.933 to 10]
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 1.5 [0.5 to 3]

11. Secondary Outcome: Population Pharmacokinetics of Dabrafenib - AUC(0-12)
Description: AUC is the area under the concentration-time curve.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
h.ng/mL
  Day 1 | 11400 (46.1)
  Day 15 | 6600 (55.6)

12. Secondary Outcome: Population Pharmacokinetics of Dabrafenib - Ctrough
Description: Ctrough is trough concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ng/mL | 77 (84.3)

13. Secondary Outcome: Population Pharmacokinetics of Dabrafenib - Racc
Description: Racc is the accumulation ratio.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Arm 1
Number analyzed (Participants) | 14
ratio | 0.624 (42.7)

14. Secondary Outcome: Population Pharmacokinetics of Hydroxydabrafenib - Cmax
Description: Cmax is the maximum peak concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 1230 (44.1)
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 1200 (58.7)

15. Secondary Outcome: Population Pharmacokinetics of Hydroxydabrafenib - Tmax
Description: Tmax is Time to Cmax (maximum peak concentration).
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Median (Full Range); unit: hr
Arm/Group | Arm 1
Number analyzed (Participants) | 20
hr
  Day 1 | 3.08 [1.45 to 10]
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 1.96 [0.967 to 3]

16. Secondary Outcome: Population Pharmacokinetics of Hydroxydabrafenib - AUC(0-12)
Description: AUC is the area under the concentration-time curve.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
h.ng/mL
  Day 1 (n=17): number analyzed (Participants) | 17
  Day 1 (n=17) | 7930 (43)
  Day 15 | 4440 (43.4)

17. Secondary Outcome: Population Pharmacokinetics of Hydroxydabrafenib - Rm/p
Description: Rm/p is the metabolite-to-parent ratio.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ratio
  Day 1 (n=17): number analyzed (Participants) | 17
  Day 1 (n=17) | 0.68 (17)
  Day 15 | 0.653 (21.4)

18. Secondary Outcome: Population Pharmacokinetics of Hydroxydabrafenib - Ctrough
Description: Ctrough is trough concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ng/mL | 94 (61.9)

19. Secondary Outcome: Population Pharmacokinetics of Hydroxydabrafenib - Racc
Description: Racc is the accumulation ratio.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Arm 1
Number analyzed (Participants) | 13
ratio | 0.56 (35.5)

20. Secondary Outcome: Population Pharmacokinetics of Desmethyl-dabrafenib - Cmax
Description: Cmax is the maximum peak concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 48.9 (93.5)
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 466 (51.6)

21. Secondary Outcome: Population Pharmacokinetics of Desmethyl-dabrafenib - Tmax
Description: Tmax is Time to Cmax (maximum peak concentration).
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Median (Full Range); unit: hr
Arm/Group | Arm 1
Number analyzed (Participants) | 20
hr
  Day 1 | 9.9 [7.92 to 10]
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 2.48 [0 to 10.1]

22. Secondary Outcome: Population Pharmacokinetics of Desmethyl-dabrafenib - AUC(0-12)
Description: AUC is the area under the concentration-time curve. AUC0-12 and Rm/p could not be calculated on Day 1 because all desmethyl-dabrafenib PK profiles on Day 1 were still ascending. Therefore, the Racc on Day 15 could not be calculated for desmethyldabrafenib.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
h.ng/mL | 3960 (52.9)

23. Secondary Outcome: Population Pharmacokinetics of Desmethyl-dabrafenib - Rm/p
Description: Rm/p is the metabolite-to-parent ratio. AUC0-12 and Rm/p could not be calculated on Day 1 because all desmethyl-dabrafenib PK profiles on Day 1 were still ascending. Therefore, the Racc on Day 15 could not be calculated for desmethyldabrafenib.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ratio | 0.616 (51.4)

24. Secondary Outcome: Population Pharmacokinetics of Desmethyl-dabrafenib - Ctrough
Description: Ctrough is trough concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ng/mL | 365 (63.7)

25. Secondary Outcome: Population Pharmacokinetics of Carboxydabrafenib - Cmax
Description: Cmax is the maximum peak concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 3760 (75.7)
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 9750 (32.8)

26. Secondary Outcome: Population Pharmacokinetics of Carboxydabrafenib - Tmax
Description: Tmax is Time to Cmax (maximum peak concentration).
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Median (Full Range); unit: hr
Arm/Group | Arm 1
Number analyzed (Participants) | 20
hr
  Day 1 | 8.94 [4 to 10.1]
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 3.5 [2 to 6.08]

27. Secondary Outcome: Population Pharmacokinetics of Carboxydabrafenib - AUC(0-12)
Description: AUC is the area under the concentration-time curve.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
h.ng/mL
  Day 1 (n=1): number analyzed (Participants) | 1
  Day 1 (n=1) | 34400 (NA) — Geometric Coefficient of Variation does not apply when n is 1
  Day 15 | 86500 (34.1)

28. Secondary Outcome: Population Pharmacokinetics of Carboxydabrafenib - Rm/p
Description: Rm/p is the metabolite-to-parent ratio.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ratio
  Day 1 (n=1): number analyzed (Participants) | 1
  Day 1 (n=1) | 3.34 (NA) — Geometric Coefficient of Variation does not apply when n is 1
  Day 15 | 12.4 (55.8)

29. Secondary Outcome: Population Pharmacokinetics of Carboxydabrafenib - Ctrough
Description: Ctrough is trough concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ng/mL | 5160 (46)

30. Secondary Outcome: Population Pharmacokinetics of Carboxydabrafenib - Racc
Description: Racc is the accumulation ratio.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Arm 1
Number analyzed (Participants) | 1
ratio | 1.51 (NA) — Geometric Coefficient of Variation does not apply when n is 1

31. Secondary Outcome: Population Pharmacokinetics of Trametinib - Cmax
Description: Cmax is the maximum peak concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 9.87 (58.1)
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 25.9 (33.3)

32. Secondary Outcome: Population Pharmacokinetics of Trametinib - Tmax
Description: Tmax is Time to Cmax (maximum peak concentration).
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Median (Full Range); unit: hr
Arm/Group | Arm 1
Number analyzed (Participants) | 20
hr
  Day 1 | 1.5 [0.483 to 4]
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 11.3 [6.64 to 17]

33. Secondary Outcome: Population Pharmacokinetics of Trametinib - AUC(0-t)
Description: Area under the concentration-time curve from time zero (predose) to last time of quantifiable concentration within a subject across all treatments
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
h.ng/mL
  Day 1 | 72.6 (27.3)
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 346 (24)

34. Secondary Outcome: Population Pharmacokinetics of Trametinib - AUC(0-24)
Description: AUC is the area under the concentration-time curve.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
h.ng/mL
  Day 1 | 72.7 (27.2)
  Day 15 (n=18): number analyzed (Participants) | 18
  Day 15 (n=18) | 357 (22.7)

35. Secondary Outcome: Population Pharmacokinetics of Trametinib - Ctrough
Description: Ctrough is trough concentration.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
ng/mL | 11.2 (25.2)

36. Secondary Outcome: Population Pharmacokinetics of Trametinib - Racc
Description: Racc is the accumulation ratio.
Time Frame: Day 1 and Day 15
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Arm 1
Number analyzed (Participants) | 15
ratio | 5.16 (15.1)

37. Post Hoc Outcome: All Collected Deaths
Description: Deaths are reported in the following categories:
  On-treatment deaths are defined as deaths that occurred after treatment start up to 30 days after study drug discontinuation.
  Post-treatment deaths are defined as deaths that occurred more than 30 days after study drug discontinuation until end of post-treatment follow up.
  Total deaths are the combination of on-treatment deaths and post-treatment deaths.
Time Frame: The collection period for mortality data occurred from start of treatment until the end of the post-treatment period, up to a maximum timeframe of 4.25 years.
Population: Safety Set (on-treatment deaths) and Full Analysis Set (total deaths)
Measure: Number; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 77
Participants
  Total Deaths | 43
  On-treatment Deaths | 16
  Post-treatment Deaths | 27

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 51 months (for both dabrafenib and also Rametinib) (approx 4.25 years).
Groups:
- All Patients: All Patients
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 16/77
Serious Adverse Events (participants affected / at risk) | 18/77
Other Adverse Events (participants affected / at risk) | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=77)
Anaemia (Blood and lymphatic system disorders) | 1
Uveitis (Eye disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Arthritis infective (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chikungunya virus infection (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Post procedural sepsis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Ejection fraction decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Confusional state (Psychiatric disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=77)
Anaemia (Blood and lymphatic system disorders) | 37
Abdominal distension (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 10
Mouth ulceration (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 18
Asthenia (General disorders) | 5
Chest discomfort (General disorders) | 4
Chest pain (General disorders) | 5
Chills (General disorders) | 15
Fatigue (General disorders) | 7
Malaise (General disorders) | 6
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 46
Cystitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 22
Alanine aminotransferase increased (Investigations) | 19
Aspartate aminotransferase increased (Investigations) | 24
Blood alkaline phosphatase increased (Investigations) | 20
Blood lactate dehydrogenase increased (Investigations) | 21
Gamma-glutamyltransferase increased (Investigations) | 6
Neutrophil count decreased (Investigations) | 29
Platelet count decreased (Investigations) | 16
Weight decreased (Investigations) | 10
Weight increased (Investigations) | 17
White blood cell count decreased (Investigations) | 35
Decreased appetite (Metabolism and nutrition disorders) | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 32
Hyperkalaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypoproteinaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 19
Headache (Nervous system disorders) | 13
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 4
Panniculitis (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 29
Skin mass (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT02083354/Prot_001.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT02083354/SAP_002.pdf